CLINICAL TRIAL: NCT03102385
Title: A Survey of Attitudes of Experienced Blood Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: New York Blood Center (Other)
Responsible Party: Principal Investigator, Christopher R. France, Ph.D., Distinguished Professor of Psychology, Ohio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-X-331
Record Dates: First submitted 2017-03-22; First posted 2017-04-05 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Blood Donors
Keywords: blood donation; motivation; donor retention
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either (1) complete an on-line motivational interview about their blood donation experience, or (2) complete an on-line knowledge interview about blood donation.
Who Masked: Participant
Masking Description: All participants were informed that they would complete an on-line interview regarding blood donation. They were not be told which of the two interviews they were completing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interview (Experimental): Complete an on-line motivational interview regarding participants' blood donation experience.
  Interventions: Behavioral: Motivational Interview
- Knowledge Interview (Placebo Comparator): Complete an on-line interview regarding participants' general knowledge about blood donation.
  Interventions: Behavioral: Knowledge Interview

INTERVENTIONS:
Behavioral: Motivational Interview — A web-based computer-tailored intervention that includes open-ended questions, reflective responses, affirmations, and summarizing, as well as informing and advising. Specific topics include 1) individual motivations for giving, 2) the relationship between past donation behavior and the individual's personal goals/values, 3) donation importance and confidence rulers, 4) addressing donor concerns, and 5) summarizing.
  Arms: Motivational Interview
Behavioral: Knowledge Interview — A web-based interview that includes open-ended questions regarding blood donation knowledge.
  Arms: Knowledge Interview

SUMMARY:
This study examines the effects of a web-based motivational interview on 1) internal motivation to donate blood; 2) donor autonomy, competence and relatedness; and 3) donation intention and behavior. The study also evaluates whether group differences in donation intention and behavior are mediated by autonomy, competence, and relatedness, and in turn, internal motivation.

DETAILED DESCRIPTION:
Voluntary blood donation is both important and necessary for the provision of a steady and safe blood supply. With an aging population and increased restrictions on who can donate blood, maintenance of a stable blood supply is essential. Although 38% of the United States population is eligible to donate, only 5% actually does so. Retention of donors is essential to assuring the continuity of a safe blood supply; repeat donors are safer, more cost effective, and less likely to experience adverse reactions. Current recruitment and retention methods may not be sufficient to encourage repeat donations. According to Self-Determination Theory, people are more likely to persist with behaviors that are internally versus externally motivated. Internal motivation is enhanced by supporting an individual's needs for autonomy, competence, and relatedness. One intervention that has shown early promise as a novel method to enhance internal motivation to donate blood is motivational interviewing. However, implementation of a motivational interviewing intervention is costly and time consuming. Given the time and money required for training and delivery of a motivational interviewing intervention, the current study is designed to test the efficacy of a newly-developed web-based version of a motivational interview. Participants will be randomly assigned to complete either an on-line motivational interview about their blood donation experience or an on-line knowledge interview about blood donation.

ELIGIBILITY:
Inclusion Criteria:

* Subject donated blood within the last week with New York Blood Center.
* Subject has made 2 or more blood donations.
* Subject is eligible to donate blood again.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1177 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Blood donation attempts | 60 weeks after index donation
  The number of blood donation attempts since their study participation will be obtained from the participants' donor records.

SECONDARY OUTCOMES:
Donation Intention | on average 1 week after index donation; on average 2 days after interview; on average 7 weeks after interview
  Intent to donate blood within the next 8 weeks will be assessed using three questions on a 7-point Likert-type scale, from 1 (disagree) to 7 (agree): I plan to donate blood in the next 8 weeks., How likely is it that you will donate blood in the next 8 weeks? and I will donate blood in the next 8 weeks. Total scores on the scale range from 3 to 21, with higher scores indicating greater intention to donate.
Donation Attitude | on average 1 week after index donation; on average 2 days after interview; on average 7 weeks after interview
  Attitudes toward blood donation will be assessed using a 6-item measure where individuals are asked to rate how donating blood in the next 8 weeks would seem using a 7-item Likert-type scale. The scale distinguishes between cognitive attitudes (evaluative judgments: useful versus useless, pointless versus worthwhile, the wrong thing to do versus the right thing to do) and affective attitudes (emotional reactions: unpleasant versus pleasant, unenjoyable versus enjoyable, frightening versus not frightening). Total scores on the scale range from 6 to 42, with higher scores reflecting more positive attitudes toward blood donation.
Donation Perceived Behavioral Control | on average 1 week after index donation; on average 2 days after interview; on average 7 weeks after interview
  Individuals' perception of control over their ability to donate blood will be assessed using a 6-item measure that assesses two components of perceived behavioral control: self-efficacy (three items) and controllability (three items). Items on the self-efficacy sub-scale ask about how confident the participant is in their ability to donate blood in the next 8 weeks, while the controllability sub-scale assesses how much control participants feel they have over whether or not they donate blood. Participants are asked to rate each item on a 7-point Likert-type scale. Total scores on the scale range from 6 to 42, with higher scores reflecting greater perception of control over ones ability to donate blood.
Donation Subjective Norms | on average 1 week after index donation; on average 2 days after interview; on average 7 weeks after interview
  Individuals' perception about subjective norms will be assessed using a six item, 7-point Likert-type scale, with anchors at 1 (disagree/unlikely) and 7 (agree/likely). Total scores on the scale range from 6 to 42. The measure assesses both descriptive norms (perceived behavior of others) and injunctive norms (what an individual believes others want from him/her).
Blood Donor Identity | on average 1 week after index donation; on average 2 days after interview; on average 7 weeks after interview
  Blood Donor Identity will be measured using an 18-item scale that examines an individual's motivation to donate on the six motivational factors proposed by Self Determination Theory: amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic regulation. Participants are asked to rate their agreement with each item on a 7-point Likert-type scale, with individual item scores ranging from 1 (not at all true) to 7 (very true). A composite score for the total scale is calculated by combining the six subscale scores using the weighting of -3, -2, -1, +1, +2, +3 for the amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic regulation subscales, respectively, in order to produce a single Relative Autonomy Index score.
Blood Donation Anxiety | on average 1 week after index donation; on average 2 days after interview; on average 7 weeks after interview
  Anxiety will be assessed using the Blood Donor Anxiety Scale, a six-item scale that assesses for both the presence (3 items) and absence (3 items) of anxiety. Participants rate their agreement on how relaxed, content, pleasant, tense, nervous and jittery they would feel if they donated blood on a 4-point scale, with anchors at 1 (not at all) and 4 (very much). Composite scores on the scale range from 3 to 12, with higher scores on the presence subscale reflecting more anxiety, and higher scores on the absence subscale reflecting less anxiety about a future donation.
Blood Donor Ambivalence | on average 1 week after index donation; on average 2 days after interview; on average 7 weeks after interview
  The 6-item ambivalence scale asks participants to rate how true a statement is for them on a 7-point scale (1=Not at all true to 7=Very true). Separate subscale scores are calculated for commitment and indecision (scores ranging from 3 to 21 for each subscale).
Psychological Need Support | on average 2 days after interview
  To assess whether the Motivational Interview intervention supported the basic psychological needs of autonomy, competence, and relatedness, a 9-item Likert-type scale will be utilized (3 items per psychological need, anchors at 1 = Not at All and 7 = Extremely).
Treatment Evaluation | on average 2 days after interview
  Participants will be asked a series of questions regarding their experience during the interview.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R France, PhD, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data may be obtained after data collection is completed. Individual participant data requests should be directed to the Principal Investigator.